CLINICAL TRIAL: NCT03872128
Title: The Role of Neuroactive Steroids in Stress, Alcohol Craving and Alcohol Use in Alcohol Use Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1608018179; 1R01AA026514-01A1 (NIH)
Record Dates: First submitted 2019-02-01; First posted 2019-03-13 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized Double-blind, placebo-controlled, parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- patients receiving 300mg PREG (Active Comparator): Patients randomly assigned to receive 300mg of pregnenolone (PREG) daily.
  Interventions: Drug: Pregnenolone300
- patients receiving 500mg PREG (Active Comparator): Patients randomly assigned to receive 500mg of pregnenolone (PREG) daily.
  Interventions: Drug: Pregnenolone500
- placebo (Placebo Comparator): Patients randomly assigned to receive a placebo daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone300 — 300mg
  Arms: patients receiving 300mg PREG
Drug: Pregnenolone500 — 500mg
  Arms: patients receiving 500mg PREG
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
To use pregnenolone (PREG; 300; 500mg) daily versus placebo (PLA) as a probe to assess the role of neuroactive steroids in individuals with alcohol use disorder (AUD).

DETAILED DESCRIPTION:
The study aims to examine the effects of PREG on a) alcohol craving, mood and neuroendocrine reactivity to brief, guided imagery exposure to stress, drug cues and neutral situations in the laboratory and b) daily alcohol intake, craving, cognition and mood in men and women with AUD; and c) sex differences in all of these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals, ages 18 to 68.
* Subjects must meet current Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-V) criteria for alcohol use disorder; documented positive urine toxicology screen for alcohol at intake or collateral information from family members, significant others, room-mates etc., on recent use.
* Subject has voluntarily given informed consent and signed the informed consent document.
* Able to read English and complete study evaluations.

Exclusion Criteria:

* Women who are pregnant, or nursing or are of childbearing potential and not practicing an effective means of birth control.
* Meet current criteria for use disorder on another psychoactive substance, such as, heroin, amphetamines, hallucinogens/Phencyclidine (PCP), excluding alcohol and nicotine.
* Any current use of opiates or past history of opiate use disorder (assessed via urine toxicology and self report).
* Current use of any psychoactive drugs (urine toxicology), including anxiolytics, naltrexone or antabuse.
* Any psychotic disorder or current Axis I psychiatric symptoms requiring specific attention.
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study.
* Hypotensive individuals with sitting blood pressure below 90/50 mmHG.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Yale Stress Center: Yale University, New Haven, Connecticut
  - Yale Stress Center, New Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Started (Participants randomized) | 30 | 30 | 31
Began Treatment | 29 | 30 | 27
Completed | 27 | 25 | 19
Not Completed | 3 | 5 | 12
Not completed — Dropped out before treatment | 1 | 0 | 4
Not completed — Lost to Follow-up | 2 | 5 | 8

BASELINE CHARACTERISTICS:
Population: Data represented here is from participants that started treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 27 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.9) | 44.8 (11.6) | 47.2 (13.3) | 46.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 31
  Male | 19 | 19 | 17 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3 | 6
  Not Hispanic or Latino | 27 | 29 | 24 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 11 | 27
  White | 17 | 20 | 12 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 27 | 86
Years of Education [Mean (Standard Deviation); unit: years] | 14 (2.3) | 14.6 (2.6) | 14.6 (2.6) | 14.4 (2.6)
Number of regular smokers [Count of Participants; unit: Participants] | 12 | 13 | 9 | 34
Years of Alcohol Use [Mean (Standard Deviation); unit: years] | 21.9 (14.9) | 17.3 (9.2) | 20 (13.5) | 19.7 (12.7)
Drinking Severity (AUDIT) [Mean (Standard Deviation); unit: score on a scale] — A screening tool designed to identify individuals who may have alcohol-related problems or alcohol use disorders (AUD). Each question is scored on a scale of 0 to 4, with a total possible score ranging from 0 to 40. Higher scores indicate a greater likelihood of alcohol-related problems or AUD.
  score on a scale | 17 (6.7) | 19.2 (7.5) | 20.3 (6.7) | 18.8 (7)
World Health Organization (WHO) Severity [Count of Participants; unit: Participants] — Number of participants [percentage of group sample] for each level of World Health Organization Severity. Cut offs have been delineated differentially for men and women. For women: Low = fewer than 1.4 drinks/day; Moderate = 2.9- >1.4 drinks/day; High = 4.3- > 2.9 drinks/day; Very High = more than 4.3 drinks/day. For men: Low = fewer than 2.9 drinks/day; Moderate = 4.3- > 2.9 drinks/day; High = 7.1- > 4.3 drinks/day; Very High = more than 7.1 drinks/day.
  Participants
    Low | 10 | 8 | 10 | 28
    Moderate | 7 | 9 | 5 | 21
    High | 6 | 6 | 6 | 18
    Very High | 6 | 7 | 6 | 19
Baseline Clinical Institute Withdrawal Assessment (CIWA) Score [Mean (Standard Deviation); unit: score on a scale] — Total score 0-67. Lower scores indicate less withdrawal symptoms.
  score on a scale | 5.1 (4.7) | 4 (4.8) | 4.8 (5.8) | 4.6 (5.1)
Lifetime Mood Disorder [Count of Participants; unit: Participants] — Number of participants endorsing a Mood Disorder based on severe combined immunodeficiency (SCID) V criteria. Possible disorders include any past diagnosis of bipolar 1 or 2, major depressive disorder, persistent depressive disorder, or other/medically induced/substance induced depressive disorder.
  Participants | 9 | 10 | 5 | 24
Lifetime Anxiety Disorder (including PTSD) [Count of Participants; unit: Participants] — Number of participants endorsing an Anxiety Disorder based on SCID V criteria.
  Participants | 9 | 9 | 10 | 28
Number of Participants Currently on Medications [Count of Participants; unit: Participants] — Stabilized on medications for treatment of medical conditions. These included peripherally acting antihypertensives, asthma, gout, diabetes. Those stabilized on antidepressants were also included.
  Participants | 17 | 15 | 14 | 46
Number of participants on depression medications [Count of Participants; unit: Participants] | 4 | 5 | 5 | 14
Total number of medical conditions [Number; unit: medical conditions] | 17 | 15 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent Drinking Days
Description: The mean percent drinking days as assessed by self report on daily smartphone monitoring and corroborated by the Substance Use Calendar over the 8 week period.
Time Frame: up to 8 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: percentage of drinking days
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
percentage of drinking days | 38.5 (5.1) | 46.6 (5.7) | 53 (6.2)
Statistical Analysis 1: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; Test type: Superiority; p = 0.009, Fisher Exact

2. Primary Outcome: Percent Heavy Drinking Days
Description: The mean percent heavy drinking days as assessed by self report on daily smartphone monitoring and corroborated by the Substance Use Calendar over the 8 week period.
Time Frame: up to 8 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
percentage of heavy drinking days | 15.2 (3.6) | 23.7 (5.1) | 22.9 (5.6)
Statistical Analysis 1: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; Test type: Superiority; p = 0.019, Fisher Exact

3. Primary Outcome: Number of Drinks Per Drinking Day
Description: Average number of drinks per drinking day as assessed by self report on daily smartphone monitoring and corroborated by the Substance Use Calendar over the 8 week period.
Time Frame: up to 8 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
drinks | 1.7 (0.3) | 2.5 (0.5) | 2.3 (0.4)
Statistical Analysis 1: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; Test type: Superiority; p = 0.044, Fisher Exact

4. Secondary Outcome: Alcohol Craving
Description: Alcohol craving assessed using the weekly Obsessive Compulsive Drinking Scale (OCDS). This 14-item scale is a quick and reliable self-rating instrument that provides a total and two subscale scores that measure some cognitive aspects of alcohol "craving". Obsessive subscale is the summation of items 1-6 with score range 0-24. Compulsive subscale is the summation of items 7-14 with score range 0-32. Total score range 0-40. Higher scores indicate more obsessions and compulsions with alcohol.
Time Frame: 8 week outcome period
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
score on a scale
  OCDS: Total | 13.8 (0.5) | 16.2 (0.6) | 20.4 (0.7)
  OCDS: Obsessive | 4 (0.2) | 5.8 (0.3) | 6.9 (0.4)
  OCDS: Compulsive | 9.8 (0.3) | 10.4 (0.4) | 13.5 (0.4)
Statistical Analysis 1: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; OCDS: Total; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; OCDS: Obsessive; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; OCDS: Compulsive; Test type: Superiority; p = 0.003, Fisher Exact

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: The Systematic Assessment of Treatment Emergent Events (SAFTEE) Questionnaire will be used to assess adverse events weekly during the trial. Data presented here is the number of participants that had any adverse events while on study.
Time Frame: up to 8 weeks
Population: Participants who were randomized and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
Participants | 10 | 9 | 8

6. Secondary Outcome: Pregnenolone Levels
Description: Mean of blood levels of study drug assessed at 3 timepoints during the trial up to 8 weeks
Time Frame: up to 8 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
ng/dL | 5.46 (0.79) | 6.21 (0.66) | 2.42 (0.4)
Statistical Analysis 1: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; Test type: Superiority; p < .0001, Fisher Exact

7. Secondary Outcome: Weekly Negative Mood and Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) will be used; it has 2 subscales (one for depression and one for anxiety) each with 7 items. It is a brief measure of generalized symptoms of anxiety and fear. Respondents indicate how they currently feel and responses are rated on a 4-point Likert scale with total score range from 0 to 21. Total scores are the sum of all items. Total scores are reported. Higher scores indicate higher levels of depression or anxiety.
Time Frame: assessed weekly, score at week 8 reported
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
Number analyzed (Participants) | 29 | 30 | 27
score on a scale
  HADS-Depression | 4.53 (0.26) | 4.85 (0.24) | 6.55 (0.35)
  HADS-Anxiety | 5.36 (0.24) | 6.49 (0.27) | 7.31 (0.32)
Statistical Analysis 1: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; HADS-Depression; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Patients Receiving 300mg PREG vs Patients Receiving 500mg PREG vs Placebo; HADS-Anxiety; Test type: Superiority; p = 0.089, Fisher Exact

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Arm/Group | Patients Receiving 300mg PREG | Patients Receiving 500mg PREG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 1/27
Other Adverse Events (participants affected / at risk) | 10/29 | 9/30 | 7/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Receiving 300mg PREG (N=29) | Patients Receiving 500mg PREG (N=30) | Placebo (N=27)
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 1 — Return to heavy drinking and had to be referred to inpatient detoxification.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Receiving 300mg PREG (N=29) | Patients Receiving 500mg PREG (N=30) | Placebo (N=27)
Headache (Nervous system disorders) | 3 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Injury, poisoning and procedural complications - Other, specif (Injury, poisoning and procedural complications) | 3 | 4 | 0 — Injury/Pain
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 1 | 2 — Stomach pain and nausea
Infections and infestations - Other, specify (Infections and infestations) | 3 | 1 | 1 — Infection and Inflammation
Immune system disorders - Other, specify (Immune system disorders) | 1 | 1 | 0 — Cold and allergies
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 2 | 0 — Menstrual cramps
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Itching
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 — Restless leg
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 | 1 — Fatigue and Depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03872128/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03872128/ICF_001.pdf